CLINICAL TRIAL: NCT03979859
Title: Double-Blind, Randomized, Placebo-Controlled Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Multiple Ascending Oral Doses Of WCK 4873 In Healthy Adult Volunteers
Brief Title: Evaluate The Safety, Tolerability and Pharmacokinetics Of Multiple Ascending Oral Doses Of WCK 4873 In Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: W 4873 02
Record Dates: First submitted 2019-04-03; First posted 2019-06-07 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Healthy
MeSH Terms: interventions — nafithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- WCK 4873 (Experimental): 200 and 400 mg tablets Dosage form : Oral tablets Doses : To be determined based on the safety, tolerability and PK results of the single dose and food effect study
  Interventions: Drug: WCK 4873
- Placebo (Placebo Comparator): Visually matching placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: WCK 4873
  Arms: WCK 4873
Drug: Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, single center, placebo-controlled, sequential cohort study in a maximum of 3 cohorts of 10 healthy male and/or female subjects each. Subjects in Cohorts 1, 2 and 3 will receive ascending multiple oral doses of WCK 4873 or matching placebo once daily on Days 1 to 7. Dosing will be conducted under fed conditions on each dosing day. The dose levels to be administered will be based on the safety, tolerability and PK results of the single dose and food effect study (W 4873 01 study; PRA-code WOE384EC-123841).

ELIGIBILITY:
Inclusion Criteria:

* BMI : 18.0-30.0 kg/m2 (Body Mass Index [BMI] [kg/m2] = Body weight [kg] Height2 [m2])
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "power-drinks"), grapefruit (juice) from 48 h prior to entry in the clinical research center until discharge
* Medical history without major pathology as judged by the Principal Investigator
* Resting supine blood pressure 90-139 (systolic) / 40-89 (diastolic) mmHg, a resting pulse rate of 40 beats per minute or higher, and showing no clinically relevant deviations as judged by the Principal Investigator
* Computerized 12-lead electrocardiogram (ECG) recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the Principal -Investigator. QTcF should be <450 ms

Exclusion Criteria:

* Previous participation in the current study
* Evidence of clinically relevant pathology
* Mental handicap
* History of Myasthenia Gravis
* History of hepatitis and/or jaundice associated with the use of any antibiotic
* Congenital prolongation of the QTc interval, ongoing proarrhythmic conditions such as uncorrected hypokalemia or hypomagnesemia, clinically significant bradycardia
* History of relevant drug and/or food allergies
* Regular/routine treatment with non-topical medications within 30 days prior to entry into the clinical research center
* Smoking within 60 days prior to drug administration and through the follow-up visit
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2013-12-05 (Actual); Study Completion 2013-12-30 (Actual)

PRIMARY OUTCOMES:
Assessing incidence of treatment emergent AEs | Day 24
  By abnormal clinical laboratory (including liver function tests) findings
Assessing incidence of treatment emergent AEs | Day 24
  By variation in physical examination
Assessing incidence of treatment emergent AEs | Day 24
  By abnormal findings in eye movement test and visual acuity test
Assessing incidence of treatment emergent AEs | Day 24
  By abnormal vital signs
Assessing incidence of treatment emergent AEs | Day 24
  variations in 12-lead electrocardiogram
Measure the pharmacokinetic parameter: Area Under Curve (AUC) | Day 10
  plasma PK parameters area under curve (AUC)
Measure the pharmacokinetic parameter-plasma PK concentration | Day 10
  Plasma concentration -Cmax
Measure the pharmacokinetic parameter- Time | Day 10
  Plasma PK parameter- Tmax
Measure the pharmacokinetic parameter- Time | Day 10
  Plasma PK parameter- T1/2